CLINICAL TRIAL: NCT03574584
Title: An Ascending Dose Trial Investigating Safety, Tolerability and Pharmacokinetics of Multiple Weekly Doses of NNC0165-1562 and Semaglutide in Subjects With Overweight or Obesity
Brief Title: A Research Study of NNC0165-1562 and Semaglutide in People Who Are Overweight or Obese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9747-4261; U1111-1191-5147 (Other: World Health Organization (WHO))
Record Dates: First submitted 2018-06-13; First posted 2018-07-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Metabolism and Nutrition Disorders; Overweight or Obesity
MeSH Terms: conditions — Nutrition Disorders; Overweight; Obesity | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Three (3) cohorts are planned. In each cohort subjects will be assigned to trial product. Subjects will be randomised in a 3:1 manner within cohorts to receive either:
  1. Semaglutide and NNC0165-1562 once weekly (9 subjects per cohort)
  2. Semaglutide and placebo once weekly (3 subjects per cohort)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Sponsor staff involved in the clinical trial is masked according to company standard procedures.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- NNC0165-1562 + Semaglutide (Experimental): Participants will receive NNC0165-1562 and semaglutide once weekly for 20 weeks.
  Interventions: Drug: NNC0165-1562; Drug: Semaglutide; Drug: Placebo (NNC0165-1562)
- Placebo (NNC0165-1562) + Semaglutide (Experimental): Participants will receive placebo (NNC0165-1562) and semaglutide once weekly for 20 weeks.
  Interventions: Drug: NNC0165-1562; Drug: Semaglutide; Drug: Placebo (NNC0165-1562)

INTERVENTIONS:
Drug: NNC0165-1562 — Participants will receive NNC0165-1562 subcutaneous (s.c., under the skin) injection(s) once-weekly for 20 weeks. The dose will be escalated over 16 weeks to a final dose level that will be maintained for 4 weeks.
Drug: Semaglutide — Participants will receive semaglutide s.c. injection(s) once-weekly for 20 weeks. The dose will be escalated over 16 weeks to a final dose level that will be maintained for 4 weeks.
Drug: Placebo (NNC0165-1562) — Participants will receive placebo (NNC0165-1562) s.c. injection(s) once-weekly for 20 weeks.

SUMMARY:
The study is investigating new medicines for weight control in people with high body weight. The study looks at how the study medicines work in the body. Participants will get semaglutide and either NNC0165-1562 or "dummy" medicine -which treatment participants get is decided by chance. Participants will get 2 injections per week for 5 months. A study nurse at the clinic will inject the medicine with a thin needle in a skin fold in the stomach. The study will last for about 7 months. Participants will have 27 visits to the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 19-55 years (both inclusive) at the time of signing informed consent.
* Body mass index (BMI) between 27.0 and 39.9 kg/sqm (both inclusive) at screening. Obesity should be due to excess adipose tissue, as judged by the investigator.

Exclusion Criteria:

* Female subjects who are of child bearing potential (pre-menopausal and not surgically sterilised) and are sexually active with male partner(s) who are not surgically sterilised (vasectomy) and are not using highly effective contraceptive methods (Pearl Index less than 1%, such as implants, injectables, oral contraceptives, intrauterine devices, diaphragm or cervical cap+spermicide) combined with a highly effective method of contraception for their male partner(s) (e.g. condom with spermicide), or are pregnant, breast-feeding or intend to become pregnant.
* Male subjects who are not surgically sterilised (vasectomy) and are sexually active with female partner(s), who are not using a highly effective method of contraception (such as condom with spermicide) combined with a highly effective method of contraception for their non-pregnant female partner(s) (Pearl Index less than 1%, such as implants, injectables, oral contraceptives, intrauterine devices, diaphragm or cervical cap+spermicide), or intend to donate sperm in the period from screening until 3 months following administration of the investigational medical product.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-07-27 (Actual); Study Completion 2019-07-27 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events (TEAEs) | Week 0-25
  Count of adverse events.

SECONDARY OUTCOMES:
AUC0-168h,1562,SS; the area under the NNC0165-1562 plasma concentration-time curve from time 0 to 168 hours at steady state | Week 19 (day 134) to week 20 (day 141)
  Measured in nmol*h/L. Measured at hours 0, 4, 8, 16, 24, 36, 48, 60 and 168 starting on day 134.
AUC0-168h,sema,SS; the area under the semaglutide plasma concentration time curve from 0 to 168 hours at steady state | Week 19 (day 134) to week 20 (day 141)
  Measured in nmol*h/L. Measured at hours 0, 4, 8, 16, 24, 36, 48, 60 and 168 starting on day 134.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Reporting Anchor and Disclosure (1452), Study Director — Novo Nordisk A/S
Locations (2):
- United States (2):
  - Novo Nordisk Investigational Site, Tempe, Arizona
  - Novo Nordisk Investigational Site, Lincoln, Nebraska

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com/sharing-results